CLINICAL TRIAL: NCT03063723
Title: Dynamic Changes of the Frequency of Classic and Inflammatory Monocytes Subsets and Natural Killer Cells in Chronic Hepatitis C Patients Treated by Direct-acting Antiviral Agents
Brief Title: Dynamic Changes of Monocytes and NK Cells of CHC Patient Treated by DAAs
Status: Completed | Type: Observational
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Gang Ning, Principal Investigator, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: Effect of DAAs on immune cells
Record Dates: First submitted 2017-02-17; First posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Chronic Hepatitis C (Disorder)
Keywords: Chronic Hepatitis C; Monocytes; Nk cells; direct-acting antiviral agents
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — ledipasvir, sofosbuvir drug combination; daclatasvir

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CHC patients: 15 treatment-naive CHC patients treated by Ledipasvir-Sofosbuvir orDaclatasvir-Sofosbuvir.
  Interventions: Drug: Ledipasvir-Sofosbuvir; Drug: Daclatasvir-Sofosbuvir
- Healthy controls: 10 Healthy controls without any treatment

INTERVENTIONS:
Drug: Ledipasvir-Sofosbuvir — 8 CHC patients were treated with Sofosbuvir (400mg, qd)/Ledipasvir (90mg, qd) for 12 weeks
  Other Names: Harvoni
  Groups: CHC patients
Drug: Daclatasvir-Sofosbuvir — 7 CHC patients were treated with Sofosbuvir (400mg, qd)/Daclatasvir (60mg,qd) for 12 weeks.
  Other Names: Daklinza
  Groups: CHC patients

SUMMARY:
Recently,surprisingly and unexpectedly increased aggressiveness and high rates of HCC recurrence (28%(16/58) and 29%(17/59), respectively) have been reported in patients who cleared HCV with DAAs after achieving a complete response to resection or local ablation within only 6 months of therapy. The authors hypothesized that the rapid eradication of HCV and control of liver inflammation would impact anti-tumoral immune control, which in turn might contribute to the neoplastic cells proliferation. Conversely, three independent prospective French cohorts failed to reveal an increased risk of HCC recurrence after DAAs treatment in CHC patients after receiving curative cancer treatments.Although the impact of DAAs treatment on the rate of HCC occurrence or recurrence still remain unclear, it would be more important to pay attention to the immunological changes of CHC patients treated with DAAs.Up to now, little was known about the immunological changes of chronic hepatitis C (CHC) patients treated with direct-acting antiviral agents (DAAs), here we try to explore the effect of antiviral treatment of CHC patients with DAAs on the frequency of monocytes, NK cells and cytokines that promote their activation.

DETAILED DESCRIPTION:
15 treatment-naive CHC patients and 10 healthy controls were recruited. Patients were examined before DAAs therapy (0w) and at weeks 4 (4w) and weeks 12 (12w) of the therapy. The percentage of monocytes,NK cells of the peripheral blood were analyzed by flow cytometry. Serum cytokines IL-12, IL-18, CXCL10, CXCL11, sCD14 and sCD163 were measured by enzyme linked immunosorbent assay.

ELIGIBILITY:
Inclusion Criteria:

* Positive serum Anti-HCV antibody or serum HCV-RNA, CHC patients without any treatment

Exclusion Criteria:

Patient has a history of clinical signs/symptoms of hepatic decompensation (Child-Pugh Grade B or C) or ascites, esophageal variceal bleeding, hepatic encephalopathy, or spontaneous bacterial peritonitis.

Patient has a history of hepatocellular carcinoma (HCC) or suspected symptoms of HCC, such as suspicious foci on imaging studies and/or serum alpha-fetoprotein (AFP)>50ng/mL.

Patient has received IFN or other immunomodulatory treatment within 52 weeks before Screening.

Patient has a medical condition that requires frequent use of systemic acyclovir or famciclovir.

Patient has a medical condition that requires frequent use of systemic corticosteroids, however topical and inhaled corticosteroids are allowed.

Patient has used hepatotoxic drugs within one month. Patient has overtaken alcohol (>40g/day) or abused illicit drugs in recent one year.

Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive urine pregnancy test.

Patients who co-infected with HAV, HBV, HDV, HEV,HIV(human immunodeficiency virus ) Patient has one or more additional known primary or secondary causes of liver disease, other than hepatitis C (e.g., alcoholism, autoimmune hepatitis).

History of malignancy of any organ system.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 15 treatment-naive CHC patients and 10 healthy controls were recruited.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Changes of the frequency of CD3-CD16+CD56+ NK cells | 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment) and 12 weeks (12 weeks after DAAs treatment)
  Measurement of the frequency of CD3-CD16+CD56+ NK cells of peripheral blood of CHC patients at 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment) and 12 weeks (12 weeks after DAAs treatment)

SECONDARY OUTCOMES:
Changes of the frequency of classic CD14++CD16- monocytes and inflammatory CD14+CD16+ monocytes. | 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment) and 12 weeks (12 weeks after DAAs treatment)
  Measurement of the frequency of classic CD14++CD16- monocytes and inflammatory CD14+CD16+ monocytes of peripheral blood of CHC patients at 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment) and 12 weeks (12 weeks after DAAs treatment).
Changes of serum levels of IL-12 | 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment) and 12 weeks (12 weeks after DAAs treatment)
  Measurement of serum levels of IL-12 of peripheral blood of CHC patients at 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment) and 12 weeks (12 weeks after DAAs treatment).
Changes of serum levels of IL-18 | 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment) and 12 weeks (12 weeks after DAAs treatment)
  Measurement of serum levels of IL-18 of peripheral blood of CHC patients at 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment) and 12 weeks (12 weeks after DAAs treatment).
Changes of serum levels of CXCL10 | 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment) and 12 weeks (12 weeks after DAAs treatment)
  Measurement of serum levels of CXCL10 of peripheral blood of CHC patients at 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment) and 12 weeks (12 weeks after DAAs treatment).
Changes of serum levels of CXCL11 | 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment) and 12 weeks (12 weeks after DAAs treatment)
  Measurement of serum levels of CXCL11 of peripheral blood of CHC patients at 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment) and 12 weeks (12 weeks after DAAs treatment).
Changes of serum levels of sCD14 | 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment) and 12 weeks (12 weeks after DAAs treatment)
  Measurement of serum levels of sCD14 of peripheral blood of CHC patients at 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment) and 12 weeks (12 weeks after DAAs treatment).
Changes of serum levels of sCD163 | 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment) and 12 weeks (12 weeks after DAAs treatment)
  Measurement of serum levels of sCD163 of peripheral blood of CHC patients at 0 week (before DAAs treatment),4 weeks (4 weeks after DAAs treatment) and 12 weeks (12 weeks after DAAs treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Liang Gao, Study Chair — Third Affiliated Hospital, Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) is not available to other researchers.

REFERENCES:
- [Derived] Ning G, Li YT, Chen YM, Zhang Y, Zeng YF, Lin CS. Dynamic Changes of the Frequency of Classic and Inflammatory Monocytes Subsets and Natural Killer Cells in Chronic Hepatitis C Patients Treated by Direct-Acting Antiviral Agents. Can J Gastroenterol Hepatol. 2017;2017:3612403. doi: 10.1155/2017/3612403. Epub 2017 May 8. PMID 28567369